CLINICAL TRIAL: NCT05163236
Title: Sensitivity of Fecal Immunochemical Test (FIT) for Colorectal Cancer (CRC) Screening and Interval Cancer Risk : a Population Based Study
Brief Title: Sensitivity of Fecal Immunochemical Test (FIT) for Colorectal Cancer (CRC) Screening
Acronym: FITBACK
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Collaborators: Registre des Tumeurs Digestives du Finistère (Other); Centre Régional de Coordination des Dépistages des Cancers Bretagne (CRCDC Bretagne) (Unknown)
Responsible Party: Sponsor
Other Study IDs: FITBACK ( 29BRC21.0147)
Record Dates: First submitted 2021-11-18; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Neoplasms Malignant; Colonoscopy; Early Detection of Cancer; Female; Mass Screening; Middle Aged; Occult Blood
Keywords: Screening; Fecal immunochemical test; survival; interval cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- CRC in excluded population: CRC diagnosed in the population excluded from screening
  Interventions: Diagnostic Test: Fecal immunochemical test (FIT) not performed
- Screen-detected colorectal cancers (SD-CRCs): CRC diagnosed after a positive fecal immunochemical test (FIT)
  Interventions: Diagnostic Test: Positive fecal immunochemical test (FIT)
- Colorectal cancers (CRCs) with delayed diagnosis: CRCs diagnosed after a positive fecal immunochemical (FIT) test, but without colonoscopy or > 2 years after a positive fecal immunochemical test
  Interventions: Diagnostic Test: Positive fecal immunochemical test (FIT)
- Fecal immunochemical test interval colorectal cancers (FIT IC): CRCs diagnosed 2 years after a negative FIT
  Interventions: Diagnostic Test: Negative fecal immunochemical test (FIT)
- colorectal cancers (CRCs) in non-responders: CRCs diagnosed in the FIT non-responders population
  Interventions: Diagnostic Test: Fecal immunochemical test (FIT) not performed
- Post-colonoscopy interval cancers: CRCs diagnosed within 5 years after a colonoscopy performed following a positive test that did not find colorectal cancer
  Interventions: Diagnostic Test: Positive fecal immunochemical test (FIT)

INTERVENTIONS:
Diagnostic Test: Positive fecal immunochemical test (FIT) — We evaluated CRCs screening campaign from January 1, 2016 to December 31, 2017, and interval cancers within two years after a negative test, and five years for post-colonoscopy interval cancers.
  Groups: Colorectal cancers (CRCs) with delayed diagnosis; Post-colonoscopy interval cancers; Screen-detected colorectal cancers (SD-CRCs)
Diagnostic Test: Negative fecal immunochemical test (FIT) — We evaluated CRCs screening campaign from January 1, 2016 to December 31, 2017, and interval cancers within two years after a negative test, and five years for post-colonoscopy interval cancers.
  Groups: Fecal immunochemical test interval colorectal cancers (FIT IC)
Diagnostic Test: Fecal immunochemical test (FIT) not performed — We evaluated CRCs screening campaign from January 1, 2016 to December 31, 2017, and interval cancers within two years after a negative test, and five years for post-colonoscopy interval cancers.
  Groups: CRC in excluded population; colorectal cancers (CRCs) in non-responders

SUMMARY:
Fecal immunochemical test (FIT) was introduced in France late 2015, FIT has better diagnostic accuracy for colorectal cancers (CRCs) than previous screening tests. Our primary objective was to evaluate the sensitivity of FIT and the proportion of interval cancer.

DETAILED DESCRIPTION:
Fecal immunochemical test (FIT) aims to detect pre-symptomatic lesions, i.e., early stage colorectal cancers (CRCs) or pre-cancerous lesions such as colonic adenomas in order to reduce CRC mortality. FIT was introduced in France late 2015, FIT has better diagnostic accuracy for CRCs than previous screening tests. Determining the incidence of post-test interval CRCs, diagnosed after a negative FIT and before the recommended date of the next test (2-year interval), allows assessment of the sensitivity of the test. The primary objective of this study was to evaluate the performance of FIT during the CRC screening campaign in the Finistère department (France) from January 1, 2016 to December 31, 2017. Its secondary objectives were the evaluation of diagnostic circumstances and their impact on treatment and survival, and risk factors for interval cancer (IC).

ELIGIBILITY:
Inclusion Criteria:

* All subjects between 50 and 77 years diagnosed with an in situ or an invasive CRC
* Inhabitants of the Finistère area
* Subjects were included by period:

  * from January 2016 to December 2017 for subjects with SD-CRC, non-responders and the excluded population
  * from January 2016 to December 2019 for subjects with FIT-ICs (2-year interval)
  * from January 2016 to December 2020 for subjects with post-colonoscopy IC
  * from January 2018 to December 2020 for subjects with delayed diagnosis

Exclusion Criteria:

* Subjects who refused to participate in the case of refusal of data collection
* Subject swith CRC other than adenocarcinoma were excluded.

Ages: 50 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study evaluated the CRC screening campaign, which took place from January 1, 2016 to December 31, 2017 in the Finistère department.
Sampling Method: Non-Probability Sample
Enrollment: 1149 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
sensitivity of the fecal immunochemical test for the detection of colorectal cancers | We evaluated CRCs screening campaign from January 1, 2016 to December 31, 2017, and interval cancers within two years after a negative test, and five years for post-colonoscopy interval cancers.
  Sensitivity = True positive / True positive + False negative = SD CRCs / SD CRCs + FIT IC

SECONDARY OUTCOMES:
Parameters affecting the sensitivity of FIT, risk factors of interval cancer | We evaluated CRCs screening campaign from January 1, 2016 to December 31, 2017, and interval cancers within two years after a negative test, and five years for post-colonoscopy interval cancers.
  Age, sex, stages, localizations, comparison by Chi2 or Fisher's test for categorical data and Student's test for quantitative data. Multivariate analysis using logistic regression.
FIT value | FIT data included its value, comprised between 10 and 200 µg haemoglobin/g faeces (analytical limits of quantification),
  FIT value, comprised between 10 and 200 µg haemoglobin/g faeces (analytical limits of quantification),
Survival | We evaluated CRCs screening campaign from January 1, 2016 to December 31, 2017, and interval cancers within two years after a negative test, and five years for post-colonoscopy interval cancers.
  Analysis of survival according to diagnostic circumstances
Treatment | We evaluated CRCs screening campaign from January 1, 2016 to December 31, 2017, and interval cancers within two years after a negative test, and five years for post-colonoscopy interval cancers.
  Analysis of treatment according to diagnostic circumstances

CONTACTS AND LOCATIONS:
Overall Officials: Michel ROBASZKIEWICZ, Study Director — University Hospital, Brest
Locations (1):
- University Hospital, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee KJ, Inoue M, Otani T, Iwasaki M, Sasazuki S, Tsugane S; Japan Public Health Center-based Prospective Study. Colorectal cancer screening using fecal occult blood test and subsequent risk of colorectal cancer: a prospective cohort study in Japan. Cancer Detect Prev. 2007;31(1):3-11. doi: 10.1016/j.cdp.2006.11.002. Epub 2007 Feb 7. PMID 17289293
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Drouillard A, Bouvier AM, Rollot F, Faivre J, Jooste V, Lepage C. Conditional net survival: Relevant prognostic information for colorectal cancer survivors. A French population-based study. Dig Liver Dis. 2015 Jul;47(7):597-601. doi: 10.1016/j.dld.2015.03.013. Epub 2015 Mar 27. PMID 25911573
- [Background] Tinmouth J, Lansdorp-Vogelaar I, Allison JE. Faecal immunochemical tests versus guaiac faecal occult blood tests: what clinicians and colorectal cancer screening programme organisers need to know. Gut. 2015 Aug;64(8):1327-37. doi: 10.1136/gutjnl-2014-308074. Epub 2015 Jun 3. PMID 26041750
- [Background] Brenner H, Tao S. Superior diagnostic performance of faecal immunochemical tests for haemoglobin in a head-to-head comparison with guaiac based faecal occult blood test among 2235 participants of screening colonoscopy. Eur J Cancer. 2013 Sep;49(14):3049-54. doi: 10.1016/j.ejca.2013.04.023. Epub 2013 May 22. PMID 23706981
- [Background] European Colorectal Cancer Screening Guidelines Working Group; von Karsa L, Patnick J, Segnan N, Atkin W, Halloran S, Lansdorp-Vogelaar I, Malila N, Minozzi S, Moss S, Quirke P, Steele RJ, Vieth M, Aabakken L, Altenhofen L, Ancelle-Park R, Antoljak N, Anttila A, Armaroli P, Arrossi S, Austoker J, Banzi R, Bellisario C, Blom J, Brenner H, Bretthauer M, Camargo Cancela M, Costamagna G, Cuzick J, Dai M, Daniel J, Dekker E, Delicata N, Ducarroz S, Erfkamp H, Espinas JA, Faivre J, Faulds Wood L, Flugelman A, Frkovic-Grazio S, Geller B, Giordano L, Grazzini G, Green J, Hamashima C, Herrmann C, Hewitson P, Hoff G, Holten I, Jover R, Kaminski MF, Kuipers EJ, Kurtinaitis J, Lambert R, Launoy G, Lee W, Leicester R, Leja M, Lieberman D, Lignini T, Lucas E, Lynge E, Madai S, Marinho J, Maucec Zakotnik J, Minoli G, Monk C, Morais A, Muwonge R, Nadel M, Neamtiu L, Peris Tuser M, Pignone M, Pox C, Primic-Zakelj M, Psaila J, Rabeneck L, Ransohoff D, Rasmussen M, Regula J, Ren J, Rennert G, Rey J, Riddell RH, Risio M, Rodrigues V, Saito H, Sauvaget C, Scharpantgen A, Schmiegel W, Senore C, Siddiqi M, Sighoko D, Smith R, Smith S, Suchanek S, Suonio E, Tong W, Tornberg S, Van Cutsem E, Vignatelli L, Villain P, Voti L, Watanabe H, Watson J, Winawer S, Young G, Zaksas V, Zappa M, Valori R. European guidelines for quality assurance in colorectal cancer screening and diagnosis: overview and introduction to the full supplement publication. Endoscopy. 2013;45(1):51-9. doi: 10.1055/s-0032-1325997. Epub 2012 Dec 4. PMID 23212726
- [Background] Ventura L, Mantellini P, Grazzini G, Castiglione G, Buzzoni C, Rubeca T, Sacchettini C, Paci E, Zappa M. The impact of immunochemical faecal occult blood testing on colorectal cancer incidence. Dig Liver Dis. 2014 Jan;46(1):82-6. doi: 10.1016/j.dld.2013.07.017. Epub 2013 Sep 4. PMID 24011791
- [Background] Lee JK, Liles EG, Bent S, Levin TR, Corley DA. Accuracy of fecal immunochemical tests for colorectal cancer: systematic review and meta-analysis. Ann Intern Med. 2014 Feb 4;160(3):171. doi: 10.7326/M13-1484. PMID 24658694
- [Background] Parra-Blanco A, Gimeno-Garcia AZ, Quintero E, Nicolas D, Moreno SG, Jimenez A, Hernandez-Guerra M, Carrillo-Palau M, Eishi Y, Lopez-Bastida J. Diagnostic accuracy of immunochemical versus guaiac faecal occult blood tests for colorectal cancer screening. J Gastroenterol. 2010 Jul;45(7):703-12. doi: 10.1007/s00535-010-0214-8. Epub 2010 Feb 17. PMID 20157748
- [Background] Chiu HM, Chen SL, Yen AM, Chiu SY, Fann JC, Lee YC, Pan SL, Wu MS, Liao CS, Chen HH, Koong SL, Chiou ST. Effectiveness of fecal immunochemical testing in reducing colorectal cancer mortality from the One Million Taiwanese Screening Program. Cancer. 2015 Sep 15;121(18):3221-9. doi: 10.1002/cncr.29462. Epub 2015 May 20. PMID 25995082
- [Background] van der Vlugt M, Grobbee EJ, Bossuyt PMM, Bos A, Bongers E, Spijker W, Kuipers EJ, Lansdorp-Vogelaar I, Spaander MCW, Dekker E. Interval Colorectal Cancer Incidence Among Subjects Undergoing Multiple Rounds of Fecal Immunochemical Testing. Gastroenterology. 2017 Aug;153(2):439-447.e2. doi: 10.1053/j.gastro.2017.05.004. Epub 2017 May 5. PMID 28483499
- [Background] van de Veerdonk W, Hoeck S, Peeters M, Van Hal G, Francart J, De Brabander I. Occurrence and characteristics of faecal immunochemical screen-detected cancers vs non-screen-detected cancers: Results from a Flemish colorectal cancer screening programme. United European Gastroenterol J. 2020 Mar;8(2):185-194. doi: 10.1177/2050640619882157. Epub 2019 Oct 3. PMID 32213071
- [Background] Portillo I, Arana-Arri E, Idigoras I, Bilbao I, Martinez-Indart L, Bujanda L, Gutierrez-Ibarluzea I. Colorectal and interval cancers of the Colorectal Cancer Screening Program in the Basque Country (Spain). World J Gastroenterol. 2017 Apr 21;23(15):2731-2742. doi: 10.3748/wjg.v23.i15.2731. PMID 28487610

DOCUMENTS (1):
  • Informed Consent Form (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT05163236/ICF_000.pdf